CLINICAL TRIAL: NCT02126774
Title: The Human Epilepsy Project
Acronym: HEP
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: The Epilepsy Study Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: 12-02865
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Focal Epilepsy
Keywords: epilepsy; focal epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- focal epilepsy: observational study

SUMMARY:
HEP is a five-year, prospective, observational study whose primary goal is to identify clinical characteristics and biomarkers predictive of disease outcome, progression, and treatment response in participants with newly treated focal epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a serious disease. It affects approximately 2.4 million Americans, with a lifetime risk estimated at 3%. More than 181,000 Americans develop epilepsy every year, and a substantial proportion has seizures that cannot be controlled by available medications. For the vast majority of patients with epilepsy, we do not understand the biological basis of their disease; we do not know whether a given anti-epileptic drug (AED) will be effective; and we cannot predict the severity of the seizure disorder, the potential emergence of co-morbidities, or the likelihood of remission.

The Human Epilepsy Project seeks to answer these unknowns by collecting high-resolution clinical information and treatment response, MRIs, EEGs, and blood and urine samples for biomarkers. A major outcome of the project is to create an open data repository of clinical information and biologic samples for future studies.

HEP may have a transformative impact on epilepsy diagnosis and treatment by identifying critical clinical features and biomarkers at the onset of epilepsy that can be used to predict outcome and guide therapy. We hope to identify subsets of patients at high risk for pharmacoresistance who may benefit from more aggressive initial therapy and earlier consideration for surgical treatment. The existence of biomarkers that predict the likelihood of disease remission would dramatically affect treatment decisions and counseling for millions of patients.

In addition to its impact on current clinical care, the data and specimens collected in HEP, including sequential neuroimaging, electrophysiology and metabolite profiles, and banked DNA for the purpose of future genomics studies, have the potential to provide new insights into the biological basis of focal epilepsy, which will advance our efforts to discover effective treatments and cures for this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Clinical seizure(s) and history consistent with focal epilepsy
* At least two confirmed spontaneous seizures, at least 24 hours apart, in the 12 months prior to enrollment
* Complete AED history prior to enrollment (with approximate dates and doses) is available (exception can be made for AEDs taken for <1 week)
* Age ≥12 years and ≤60 years at time of seizure onset
* Age ≥12 years and ≤60 years at time of enrollment
* Treatment instituted not more than 4 months prior to enrollment
* One of the following:

  1. Normal MRI with inter-ictal EEG showing focal abnormality (focal sharp waves or focal slowing)
  2. Normal MRI and normal inter-ictal EEG, with clinical or electrographic seizure activity on ictal EEG
  3. Definitive clinical history of recurrent seizures consistent with focal epilepsy, adjudicated by central reviewers, if normal MRI and normal EEG
  4. Focal lesion (non-progressive) on MRI with normal EEG (acceptable focal lesions include MTS, FCD, single cavernoma, and AVMs that are not of large size and lack significant amounts of hemosiderin)

Exclusion Criteria:

* Idiopathic or symptomatic generalized epilepsy
* Any epilepsy etiology that could produce significant gliosis or brain injury and would be likely to alter biomarkers. These include:

  1. Epilepsy with an etiology occurring in the previous two years that would produce significant CNS injury (e.g., traumatic brain injury that involves direct disruption of brain tissue, stroke, encephalitis)
  2. History of intracranial bleeding (e.g., subarachnoid, intraparenchymal)
* Identified genetic epilepsy syndrome
* Presence of moderate or greater developmental or cognitive delay prior to seizure onset (e.g., if an adolescent, not in self-contained classroom; if IQ is documented, should be > 70)
* History of chronic drug or alcohol abuse within the last 2 years
* IGE/focal epilepsy mixed syndromes
* Progressive neurological disorder (brain tumor, AD, PME, etc.)
* Major medical co-morbidities such as renal failure requiring dialysis, metastatic cancer, HIV, or significant liver or renal disease
* Autism Spectrum Disorder
* Seizures only during pregnancy
* History of previous or current significant psychiatric disorder that would interfere with conduct of the study

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Epilepsy/Neurology clinical centers
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Presence of Biomarker(s) Predictive of Anti-epileptic Drug Treatment Response | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Kuzniecky, MD, Principal Investigator — New York University, Comprehensive Epilepsy Center; Jacqueline French, MD, Principal Investigator — New York University, Comprehensive Epilepsy Center; Daniel Lowenstein, MD, Principal Investigator — University of California, San Francisco, Department of Neurology
Locations (30):
- United States (26):
  - University of Alabama, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - North Shore-LIJ Health System, Great Neck, New York
  - Albert Einstein College of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, Houston, Texas
- Australia (3):
  - Austin Hospital, University of Melbourne, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - Prince of Wales Hospital, University of New South Wales, Sydney
- University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Barnard SN, Chen Z, Holmes M, Kanner AM, Hegde M, Kuzniecky R, Lowenstein D, French JA; Human Epilepsy Project (1) Investigators. Treatment Response to Antiseizure Medications in People With Newly Diagnosed Focal Epilepsy. JAMA Neurol. 2025 Oct 1;82(10):1022-1030. doi: 10.1001/jamaneurol.2025.2949. PMID 40853673
- See also: HEP website — http://humanepilepsyproject.org